CLINICAL TRIAL: NCT03437811
Title: Efficacy of Med Systems' Electro Flo Percussor Model 5000, Airway Clearance System, for Pulmonary Clearance of Secretions.
Brief Title: Airway Clearance System (K031876) Phase IV Device Efficacy
Status: Completed | Type: Observational
Sponsor: Mack Biotech, Corp. (Industry)
Responsible Party: Principal Investigator, Leigh J. Mack, Principal Investigator (CEO), Mack Biotech, Corp.
Other Study IDs: 201801MEDSystems
Record Dates: First submitted 2018-01-17; First posted 2018-02-19 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Cystic Fibrosis, Pulmonary
Keywords: airway clearance system; cystic fibrosis; lung secretion clearance
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Active Treatment: Active arm, Electro Flo Percussor, Model 5000 airway clearance system for daily basis as needed (pro re nata).
  Interventions: Device: Electro Flo Percussor, Model 5000

INTERVENTIONS:
Device: Electro Flo Percussor, Model 5000 — FDA 510K K031876 Regulation Number: 21 CFR 868.5665 Regulation Name: Percussor, Powered-Electric Regulation Class: II Product Code: BY1

SUMMARY:
Phase IV interventional study of adults (18 to 55) having a diagnosis of cystic fibrosis (mild, moderate or severe). The study is completely voluntary and is designed to measure participants use and the effectiveness of the device within the 510K indication of: airway clearance therapy when external manipulation of the thorax. The trial period shall be 21 days and include use of a FDA cleared pulse oximetry monitor (K131111), manual spirometer as well as completion of semi-weekly participant survey.

DETAILED DESCRIPTION:
Phase IV interventional study, of participants with cystic fibrosis with mild, moderate or severe conditions, for the efficacy of the Electro Flo Percussor, Model 5000 (K031876), Regulation Number: 21 CFR 868.5665, with current FDA indication of: provide airway clearance therapy when external manipulation of the thorax is the physician's choice of treatment. Indications for this form of therapy are described by the American Association for Respiratory Care (AARC) in the Clinical Practices Guidelines for Postural Drainage Therapy ( I ) (1991). According to AARC guidelines, specific indications for external manipulation of the thorax include evidence or a suggestion of retained secretions, evidence that the patient is having difficulty with the secretion clearance, or presence of atelectasis caused by mucus plugging. In addition, the Med Systems Electro Flo Percussor Model 5000 is also indicated for external manipulation of the thorax to promote airway clearance or improve bronchial drainage for purposes of collecting mucus for diagnostic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with cystic fibrosis (mild, moderate or severe)
* Prescribed (licensed medical provider) airway clearance device/system for at home, self-treatment for airway clearance
* Physically able to perform self-treatment or treatment by an at home medical provider

Exclusion Criteria:

* History of tobacco use
* History of excessive alcohol consumption, more than 2 drinks per day, 10 per week
* Any other medical condition that would preclude use of an airway clearance device
* Previously diagnosed with major cardiological disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 18 to 55 years of age, male or female.non-smokers
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Percentage change of oxygen levels in the blood (pulse oximetry). | Change from baseline up to 3.5 hours.
  SpO2 will be monitored using the standard pulse oximeter system (K131111).

SECONDARY OUTCOMES:
Percentage change of lung function | Change from baseline up to 3.5 hours
  Evaluate expiratory forced vital capacity (FVC) and forced expiratory volume (FEV1) will be monitored with standard spirometer.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh J Mack, MD, PhD, CPI, Principal Investigator — Mack Biotech, Corp.
Locations (1):
- MED Systems, Inc., San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Available final outcomes for complete study shall be available December 31, 2019. No individual specific outcomes shall be shared.

REFERENCES:
- [Background] Main E, Prasad A, Schans C. Conventional chest physiotherapy compared to other airway clearance techniques for cystic fibrosis. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD002011. doi: 10.1002/14651858.CD002011.pub2. PMID 15674888
- [Background] Oermann CM, Sockrider MM, Giles D, Sontag MK, Accurso FJ, Castile RG. Comparison of high-frequency chest wall oscillation and oscillating positive expiratory pressure in the home management of cystic fibrosis: a pilot study. Pediatr Pulmonol. 2001 Nov;32(5):372-7. doi: 10.1002/ppul.1146. PMID 11596162
- See also: Cleared device information — http://www.medsystems.com/products/electro-flo-5000/

DOCUMENTS (3):
  • Statistical Analysis Plan (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT03437811/SAP_001.pdf
  • Study Protocol (2018-12-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT03437811/Prot_003.pdf
  • Informed Consent Form (2018-12-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT03437811/ICF_004.pdf